CLINICAL TRIAL: NCT04319445
Title: Mindfulness During COVID-19 - Remote Mindfulness Sessions
Brief Title: Mindfulness During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00064587
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-03

CONDITIONS: Migraine Disorders; Stress; Anxiety
Keywords: COVID-19
MeSH Terms: conditions — Migraine Disorders; Anxiety Disorders; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Migraine Patients/Providers/Faculty/Staff/Other (Experimental)
  Interventions: Behavioral: Mindfulness session(s)

INTERVENTIONS:
Behavioral: Mindfulness session(s) — The sessions will be hosted online using an online platform (such as through webex, private YouTube page, Facebook live, etc).

SUMMARY:
The objective of this study is to provide remote mindfulness session(s) to help during the COVID-19 pandemic.

DETAILED DESCRIPTION:
The objective of this study is to provide remote mindfulness session(s) to help during the COVID-19 pandemic.The investigators are interested in targeting patients with migraine, providers, faculty and staff. The investigators are hopeful that this will positively impact overall well-being at this stressful time. The investigators are interested in assessing feasibility, accessibility, and overall interest of an online mindfulness intervention in these populations at this time.

ELIGIBILITY:
Inclusion Criteria:

* Any person interested in participating in the mindfulness session will be eligible to complete the pre/post surveys and participate in the mindfulness session.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Wells, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Started | 144
Completed | 144
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 108
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 144

OUTCOME MEASURES:

1. Primary Outcome: Helpfulness of the Session
Description: Percentage of Participants who Felt the Mindfulness Session was Helpful - After the mindfulness session, participants used a Likert scale rating to respond to the question "How helpful was this session for you?"
Time Frame: Post-Intervention (upon completion of session up to 15 minutes)
Measure: Number; unit: percentage of participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
percentage of participants | 89

2. Primary Outcome: Platform Effectiveness
Description: Percentage of Participants who Perceived the Electronic Platform to be Effective for Practicing Mindfulness - After the mindfulness session, participants used a Likert scale rating to respond to the question "Did you find this electronic platform effective for practicing mindfulness?"
Time Frame: Post-Intervention (upon completion of session up to 15 minutes)
Measure: Number; unit: percentage of participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
percentage of participants | 89

3. Secondary Outcome: Change in Anxiety Level
Description: Percentage of Participants With Reduction in Anxiety After Mindfulness Session - Before and after the mindfulness session, participants responded to the question, "At this moment, how anxious do you feel?"
Time Frame: Pre- Intervention, Post-Intervention (upon completion of session up to 15 minutes)
Measure: Number; unit: percentage of participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
percentage of participants | 76

4. Secondary Outcome: Change in Stress Level
Description: Percentage of Participants With Reduction in Stress After Mindfulness Session - Before and after the mindfulness session, participants responded to the question, "At this moment, how much stress do you feel?"
Time Frame: Pre- Intervention, Post-Intervention (upon completion of session up to 15 minutes)
Measure: Number; unit: percentage of participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
percentage of participants | 80

5. Secondary Outcome: Value of the Session
Description: Percentage of Participants who Felt the Mindfulness Session was Valuable - After the mindfulness session, participants used a Likert scale rating to respond to the question "How much was the session of value to you?"
Time Frame: Post-Intervention (upon completion of session up to 15 minutes)
Measure: Number; unit: percentage of participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
percentage of participants | 87

6. Secondary Outcome: Satisfaction With the Session
Description: Percentage of Participants who were Satisfied with the Mindfulness Session - After the mindfulness session, participants used a Likert scale rating to respond to the question "How satisfied are you with this experience?"
Time Frame: Post-Intervention (upon completion of session up to 15 minutes)
Measure: Number; unit: percentage of participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
percentage of participants | 92

7. Secondary Outcome: Percentage of Participants That Showed Interest in a Future Session
Description: Percentage of participants that showed interest in a future session
Time Frame: Post-Intervention (upon completion of session up to 15 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
Participants | 131

8. Secondary Outcome: Percentage of Participants That Would Recommend This Session to a Family Member
Description: Percentage of participants that would recommend this session to a family member
Time Frame: Post-Intervention (upon completion of session up to 15 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
Participants | 137

9. Secondary Outcome: Percentage of Participants by Session Frequency Preference - Daily
Description: Percentage of participants that would prefer to participate in daily similar sessions again if offered
Time Frame: Post-Intervention (upon completion of session up to 15 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
Participants | 51

10. Other Pre Specified Outcome: Decreased Concern Level About the COVID 19 Pandemic
Description: Percent of Participants With Reduction in Concern over COVID-19 After Mindfulness Session - Before and after the mindfulness session, participants responded to the question, "At this moment, how concerned are you about the Coronavirus pandemic?"
Time Frame: Pre- Intervention, Post-Intervention (upon completion of session up to 15 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
Participants | 79

11. Secondary Outcome: Percentage of Participants by Session Frequency Preference - Weekly
Description: Percentage of participants that would prefer to participate in weekly similar sessions again if offered
Time Frame: Post-Intervention (upon completion of session up to 15 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
Participants | 69

12. Secondary Outcome: Percentage of Participants by Session Frequency Preference - Monthly
Description: Percentage of participants that would prefer to participate in monthly similar sessions again if offered
Time Frame: Post-Intervention (upon completion of session up to 15 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
Number analyzed (Participants) | 144
Participants | 24

ADVERSE EVENTS:
Time Frame: 15 minutes
Arm/Group | Migraine Patients/Providers/Faculty/Staff/Other
All-Cause Mortality (participants affected / at risk) | 0/144
Serious Adverse Events (participants affected / at risk) | 0/144
Other Adverse Events (participants affected / at risk) | 0/144

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT04319445/Prot_001.pdf
  • Informed Consent Form (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT04319445/ICF_000.pdf